CLINICAL TRIAL: NCT01097681
Title: An Open-Label Study to Assess the Effect of Different Grades of Renal Impairment in Japanese Patients With Type 2 Diabetes Mellitus on the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of ASP1941 Relative to Type 2 Diabetes Mellitus Patients With Normal Renal Function
Brief Title: A Study to Assess the Pharmacokinetics, Pharmacodynamics of ASP1941 in Diabetes Mellitus Patients With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1941-CL-0073
Record Dates: First submitted 2010-03-31; First posted 2010-04-02 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Urinary glucose excretion; Diabetes mellitus; ASP1941
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — ipragliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal renal function group (Experimental): oral
  Interventions: Drug: ASP1941
- Mild renal impairment group (Experimental): oral
  Interventions: Drug: ASP1941
- Moderate renal impairment group (Experimental): oral
  Interventions: Drug: ASP1941

INTERVENTIONS:
Drug: ASP1941 — oral

SUMMARY:
The primary objective of this study is to compare the pharmacokinetics of ASP1941 in type 2 diabetes mellitus patients with normal renal function and those with mild or moderate renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients for at least 12 weeks
* Fasting plasma glucose level of < 240 mg/dL
* Body Mass Index ( BMI )20.0 - 35.0kg/m2
* GFR value based on the Japanese GFR estimation equation at screening, of ≥ 30 ml/min/1.73m2

Exclusion Criteria:

* Type 1 diabetes mellitus patients
* Receiving insulin within 12 weeks before screening
* Diabetic ketoacidosis
* Dysuria and/or urinary tract infection, genital infection
* Significant renal, hepatic or cardiovascular diseases
* Severe gastrointestinal diseases

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-02-16 (Actual); Primary Completion 2010-06-18 (Actual); Study Completion 2010-06-18 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of ASP1941 | For 72 hours after dosing

SECONDARY OUTCOMES:
Urinary levels of ASP1941 | For 72 hours after dosing
Urinary glucose excretion | For 72 hours after dosing
Safety assessed by adverse events, vital signs, laboratory tests and 12-lead ECGs | For 72 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (2):
- Japan (2):
  - Kansai
  - Kantou

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results Web site — https://astellasclinicalstudyresults.com/study.aspx?ID=92